CLINICAL TRIAL: NCT03318913
Title: Effect of Acute Fish Protein Hydrolysates Ingestion on Vascular Function of the Type 2 Diabetes Subjects
Brief Title: Vascular Function, Fish Protein Hydrolysates and Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Thiago Alvares, D.sc, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 53392216.0.0000.5699
Record Dates: First submitted 2017-10-18; First posted 2017-10-24 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Vascular function; Type 2 diabetes mellitus; Fish protein hydrolysates
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Health control (No Intervention): Health young subjects free of diabetes mellitus and nutritional intervention
- DM Placebo (Placebo Comparator): Sucralose
  Interventions: Other: Placebo
- DM FHP (Active Comparator): Fish protein hydrolysates
  Interventions: Other: Fish protein hydrolysates

INTERVENTIONS:
Other: Placebo — 5g of the sucralose administered as white plastic capsules
  Arms: DM Placebo
Other: Fish protein hydrolysates — 5g of the FPH dissolving in 100 mL of water
  Arms: DM FHP

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a chronic metabolic disease of abnormal carbohydrate metabolism which is related with high morbidity and mortality rates caused by its complications. One of the major diabetes-related arterial phenotypes thought to be responsible for development of cardiovascular disease is endothelial dysfunction. Nitric oxide (NO) is a potent molecule derived of endothelium, which plays key role in control of vascular tone. In T2DM present endothelial dysfunction due to reduced NO bioavailability. Fish protein hydrolysates (FPH) have been showed to present antioxidant peptides (and high value of ACE inhibition activity. Therefore, the present study aimed to examine whether single dose of FPH ingestion would reversal macro- and microvascular endothelial dysfunction in T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus

Exclusion Criteria:

* History of symptomatic coronary artery disease;
* Stroke or other known atherosclerotic disease;
* Cancer;
* HIV positive;
* Alcohol or drug abuse within the past 6 months previous the visit 1;
* use any antioxidant supplementation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation | 60 min after nutritional intervention
  macrovascular endothelial function
Near infrared spectroscopy | 70 min after nutritional intervention
  microvascular endothelial function
High performance liquid chromatography | 75 min after nutritional intervention
  serum amino acids

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio de Janeiro, Macaé, Rio de Janeiro, Brazil